CLINICAL TRIAL: NCT02348684
Title: Pilot Study to Evaluate Cardiac Function Using Cardiac MRI and Dosimetric Correlation in Women Treated for Node Positive Breast Cancer With Three- Dimensional Conformal Radiation Therapy (3DCRT)
Brief Title: Evaluate Cardiac Function Using Cardiac MRI and Dosimetric Correlation
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Carmen Bergom, Associate Professor, Medical College of Wisconsin
Other Study IDs: Cardiac MRI post RT Breast Ca
Record Dates: First submitted 2014-08-22; First posted 2015-01-28 (Estimated); Results first posted 2019-07-01 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Node Positive Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Radiation therapy groups: Risk groups based on dosimetric radiation parameters.
  Interventions: Radiation: Radiation therapy groups

INTERVENTIONS:
Radiation: Radiation therapy groups — Radiation Therapy treatment between 2000 and 2007.
  Other Names: Regional nodal irradiation following lumpectomy/mastectomy.

SUMMARY:
The association between radiation exposure and cardiac disease is well recognized, it is not fully understood if there exists an optimal or "safe" radiation dose-volume relationship.

DETAILED DESCRIPTION:
Identification of "safe" dose volume constraints (DVC) for the heart from breast cancer radiotherapy would permit maximal oncologic benefit from radiation, identifying which patients require more complicated and resource consumptive radiation methods such as respiratory-gating or intensity modulated radiotherapy (IMRT) and establish patients who need targeted follow-up for their long term cardiac risk. Two recent technical developments now make it conceivable to identify the dose-volume relationship between heart dose and subsequent cardiac event risk: 1. CT based three dimensional conformal radiation delivery methods (3DCRT) where the precise radiation dose to any given heart volume is known, and 2. Cardiac MRI (CMR) that is more sensitive to prior methods of cardiac evaluation (e.g. SPECT) for detecting and measuring cardiac injury.

An MRI, subject health questionnaire, clinical and dosimetric data will be included in the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Women with node positive breast cancer treated with surgery, anthracycline-based or similar cardiotoxic chemotherapy, and regional nodal irradiation between 2000-2007.

Exclusion Criteria:

* Women who have not received anthracycline-based or similar cardiotoxic chemotherapy, and regional nodal irradiation between 2000-2007.

Ages: 18 Years to 95 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women Treated for Node Positive Breast Cancer with Three-Dimensional Conformal Radiation Therapy (3DCRT)
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-03; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carmen R Bergom, MD, PhD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Data available upon request after publication of findings.

REFERENCES:
- [Background] Assomull RG, Prasad SK, Lyne J, Smith G, Burman ED, Khan M, Sheppard MN, Poole-Wilson PA, Pennell DJ. Cardiovascular magnetic resonance, fibrosis, and prognosis in dilated cardiomyopathy. J Am Coll Cardiol. 2006 Nov 21;48(10):1977-85. doi: 10.1016/j.jacc.2006.07.049. Epub 2006 Oct 31. PMID 17112987

RESULTS

PARTICIPANT FLOW:
Groups:
- Radiation Therapy Groups: Risk groups based on dosimetric radiation parameters and eligibility criteria.
  Radiation therapy groups: 3D Conformal Radiation Therapy (3DCRT) to breast/chestwall and regional lymph nodes with treatment between 2000 and 2009.
Period: Overall Study
Arm/Group | Radiation Therapy Groups
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Radiation Therapy Groups
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Cardiac MRI Parameters
Description: Cardiac MRI parameters include Left Ventricular (LV) ejection fraction, LV mass (indexed), LV dimensions, extracellular volume (ECV), and late gadolinium enhancement (LGE).
Time Frame: day of MRI scan
Measure: Number; unit: number of patients
Groups:
- Radiation Therapy Groups: Risk groups based on dosimetric radiation parameters and eligibility criteria.
  Radiation therapy groups: Radiation Therapy treatment between 2000 and 2009.
Arm/Group | Radiation Therapy Groups
Number analyzed (Participants) | 20
number of patients
  LGE | 0
  LVEF, more than 1% outside normal range | 0
  LV mass (indexed), higher than normal | 0
  LV chamber dimensions, higher than normal | 0
  Total Myocardial ECV, above 30% | 3

2. Secondary Outcome: Correlate Cardiac MRI Parameters
Description: Correlate cardiac MRI parameters with pre-treatment heart imaging and cardiac dose volume constraints as a measure of cardiac injury after partial heart irradiation in women with node positive breast cancer treated with surgery, anthracycline-based chemotherapy and regional nodal irradiation.
Time Frame: the day of MRI
Reporting Status: Not Posted, anticipated posting 2021-12

3. Other Pre Specified Outcome: Dose-volume Constraints for the Heart During Radiation Therapy for Breast Cancer.
Description: Trial data will improve the understanding of cardiac function after radiotherapy and allow oncologists to start to define safe dose-volume constraints for the heart in women treated with regional nodal irradiation for breast cancer.
Time Frame: The day of the MRI
Reporting Status: Not Posted, anticipated posting 2021-12

ADVERSE EVENTS:
Arm/Group | Radiation Therapy Groups
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes